CLINICAL TRIAL: NCT06651359
Title: Development and Preliminary Evaluation of a Tailored mHealth App Designed to Improve Quality-of-Life Outcomes in Ethnically-Diverse Black Prostate Cancer Survivors (SAFE-CaPs)
Brief Title: Using a mHealth App to Improve Quality-of-Life Outcomes in Black Prostate Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OU202403MA-MHEALTH; PC230551 (Other Grant/Funding Number: DoD CDMRP PCRP)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: mHealth; Black men; Black survivors; native-born Black man; African-born Black man; Caribbeanborn Black man
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants in this arm will be eligible Black men who have prostate cancer and are either currently undergoing treatment or are cancer survivors.
  Interventions: Behavioral: Surveys for Quality of Life
- Intervention group (Experimental): Participants in this arm will be eligible Black men who have prostate cancer and are either currently undergoing treatment or are cancer survivors, who are given access to the mHealth app for this study.
  Interventions: Behavioral: Surveys for Quality of Life; Behavioral: Surveys and mHealth App access

INTERVENTIONS:
Behavioral: Surveys for Quality of Life — This group will take scheduled electronic surveys (at the beginning of the study, months 3, 6, 9, and 12) to assess the overall impact of prostate cancer on quality of life (QoL).
Behavioral: Surveys and mHealth App access — This group will take scheduled electronic surveys (at the beginning of the study, months 3, 6, 9, and 12) to assess the overall impact of prostate cancer on quality of life (QoL). Additionally, they will have a brief "initial study visit," in-person or virtually, to review the app use. This arm of participants will use the mobile application at home for 12 months. During the first 12 weeks, the application will send daily surveys about symptoms, dietary and physical activities, weekly surveys about their mood, and an assessment of their overall QoL every 3 months. The app will provide tailored educational content, including short readings, videos, and audio recordings, to help users learn more about managing symptoms and improving their functioning. After 12 months of app use, an interview will be conducted to gather feedback about their experiences with the app. The information collected from these interviews will be analyzed to further enhance and improve the app's functionality.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to ensure that the mobile health application for Black patients with prostate cancer (either actively undergoing treatment or survivors) is usable and acceptable to patients, get feedback about how to improve the app and assess its usefulness in examining their quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a culturally appropriate and specific mobile app for ethnically diverse Black men with prostate cancer (either those actively undergoing treatment or survivors) to empower them to be active participants in their care. This app will provide 1) relevant information/education about prostate cancer-specific to Black men; 2) symptoms monitoring - allowing participants to report difficulties and prompting providers to respond to concerns; and 3) testimonials from other patients with shared experiences.

All participants will be asked to complete surveys online when they start and then again at 3, 6, 9, and 12 months. A subset of randomized participants will be provided access to this app, which they will be asked to use at home for 12 months. The app users will answer daily surveys about their symptoms and activities as well as weekly mood assessments for 3 months. At the end of the 12 months, interviews will be conducted to receive feedback regarding the app.

ELIGIBILITY:
Inclusion Criteria:

- Ethnically-diverse Black prostate cancer (CaP) survivors who are either native-born, Caribbean-born, or African-born, within the early phase of their CaP survivorship journey (defined as within the first five years after diagnosis).

Exclusion Criteria:

* Men from other races.
* Men who have never been diagnosed with CaP
* Men who have the inability to speak English
* Men who do not own a smartphone
* Black CaP survivors who are over 5 years since the time of diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-08-24 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Overall Quality of Life (QoL) assessment in Black men with prostate cancer | 12 months
  The proportion of patients in the intervention arm reporting increased QoL using the Functional Assessment of Cancer Therapy - Prostate (FACT-P) survey.
  FACT-P has five subscales:
  1. Physical Well-Being- Evaluate symptoms like pain and energy.
  2. Social/Family Well-Being- Measures support and communication satisfaction.
  3. Emotional Well-Being- Assesses sadness, anxiety, coping, and hope.
  4. Functional Well-Being- Measures daily activities, contentment, and enjoyment.
  5. Prostate Cancer Subscale- Addresses symptoms like sexual function, pain, and urinary issues.
  Higher scores indicating better QoL overall. FACT-P captures physical, social, emotional, functional, and prostate-specific well-being to measure comprehensive patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Motolani Adedipe, PhD, DPh, MS, Principal Investigator — University of Oklahoma
Locations (3):
- United States (3):
  - Florida State University, Tallahassee, Florida
  - Georgia College & State University, Milledgeville, Georgia
  - University of Oklahoma HSC, Oklahoma City, Oklahoma